CLINICAL TRIAL: NCT07158645
Title: A Study to Assess Human Pharmacokinetics of a Medical Food Containing Tri-betahydroxybutyrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroEnergy Ventures, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BIO-1708
Record Dates: First submitted 2025-08-06; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: pK Study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20gTri-betahydroxybutyrin (Active Comparator): Medical Food Containing 20g Tri-betahydroxybutyrin
  Interventions: Other: Medical Food Tri-betahydroxybutyrin
- 40g Tri-betahydroxybutyrin (Active Comparator): Medical Food Containing 40g Tri-betahydroxybutyrin
  Interventions: Other: Medical Food Tri-betahydroxybutyrin
- 60g Tri-betahydroxybutyrin (Active Comparator): Medical Food Containing 60g Tri-betahydroxybutyrin
  Interventions: Other: Medical Food Tri-betahydroxybutyrin

INTERVENTIONS:
Other: Medical Food Tri-betahydroxybutyrin — Medical Food Containing Tri-betahydroxybutyrin
  Other Names: Medical Food Containing Tri-betahydroxybutyrin

SUMMARY:
The objective of this clinical trial is to obtain PK information following the acute intake of a medical food containing tri-betahydroxybutyrin (3BHB) in 18 healthy male subjects. Blood samples will be obtained for the PK analysis of beta-hydroxybutyrate and acetoacetate at t = 1 and 2 h ± 5 min, where t = 0 h is the start of study product consumption. Subjects will be administered a standard breakfast immediately following the t = 2 h blood draw. Subjects will consume the breakfast meal within 30 min and will be instructed to eat until comfortably full.

Blood samples will be obtained via the indwelling venous catheter or venipuncture at t = 3, 4, 6, 8, and 12 h ± 5 min, where t = 0 h is the start of study product consumption, for the PK analysis of beta-hydroxybutyrate and acetoacetate. Subjects will be administered a standard snack (immediately following the t = 4 h blood draw), a standard lunch (immediately following the t = 6 h blood draw) and a standard dinner (at t = 10 h) Subjects will consume the meals/snack within 30 min and will be instructed to eat until comfortably full. Following the final blood draw of Visit 2 (day 0) at t = 12 h ± 5 min, the catheter will be removed, AEs will be assessed and a standard snack will be administered for consumption prior to discharge from the clinic.

At Visit 3 (day 1), subjects will return to the clinic for clinic visit procedures (i.e., vital signs; review inclusion and exclusion criteria for relevant changes, and concomitant medication/supplement use review). AEs will be assessed and subjects will be queried about study instructions compliance. Blood samples will be obtained at t = 24 h ± 5 min (with backups) by venipuncture for the PK analysis of beta-hydroxybutyrate and acetoacetate, where t = 0 h is the time of study product consumption.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is a generally healthy male at least 60 years of age.

  2. Subject has at least a high school diploma or the equivalent.

  3. Subject has a score of 7 to 10 on the Vein Access Scale at Visit 1 (day -7).

  4. Subject has a BMI of 18.5 and 29.9 kg/m2, inclusive at Visit 1 (day -7).

  5. Subject is willing to remain on a stable dose of prescription medications within 30 d prior to Visit 1 (day -7) and throughout the study period.

  6. Subject is willing to avoid alcohol and intentional exercise 24 h prior to Visit 2 (day 0) and throughout the study period.

  7. Subject is willing to maintain habitual diet, physical activity patterns, and body weight throughout the trial.

  8. Subject is willing and able to comfortably abstain from caffeine prior to (10-14 h, target 12 h) and throughout the duration of all clinic visits (up to 14 h on Visit 2; day 0). (This is not a threat to validity to cognitive function; only possible alertness.)

  9. Subject is a non-user of all tobacco, smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches) within 6 months of Visit 1 (day -7) and has no plans to change status during the study period.

  10. Subject is willing and able to comply with the visit schedule.

  11. Subject has no health conditions that would prevent him from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history, physical examination findings, and routine laboratory test results.

  12. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Subject is female.
2. Subject has a fasting glucose greater than 125 mg/dL at Visit 1 (day -7). No retest allowed.
3. Subject has abnormal laboratory test results of clinical significance at Visit 1 (day -7) on the basis of age and gender specific reference values and/or at the discretion of the Clinical Investigator, who has MD qualifications. One re-test will be allowed on a separate day prior to Visit 2 (day 0), for subjects with abnormal laboratory test results.
4. Subject has a known allergy or sensitivity to any of the ingredients in the study products and/or any ingredients of the meals provided.
5. Subject has any signs or symptoms of an active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 d prior to Visit 2 (day 0). If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved (at the discretion of the Clinical Investigator) and any treatment (e.g., antibiotic therapy) has been completed at least 5 d prior to testing.
6. Subject experiences evidence of delirium, confusion, or other disturbances of consciousness.
7. Subject has a history of diagnosed depression in the prior 2 years of Visit 1 (day -7).
8. Subject has any diagnosed neurologic disorder that could produce cognitive deterioration including, but not limited to, Alzheimer's disease, Parkinson's disease, stroke, intracranial hemorrhage, local brain lesions including tumors, and normal pressure hydrocephalus.
9. Subject has a history of any infective or inflammatory brain disease, including those of viral, fungal, or syphilitic etiologies.
10. Subject has a history of repeated minor head injury (e.g., in boxing) or a single injury resulting in a period of unconsciousness for 1 h or more.
11. Subject has a history or presence of any acutely unstable medical condition, behavioral, and/or psychiatric disorder or surgical history that could affect the safety of the subject or interfere with study efficacy, safety, PK assessments, or the ability of the subject to complete the trial per the judgment of the Clinical Investigator (has MD qualifications).
12. Subject has a history or presence of clinically important endocrine (including hyperparathyroidism, type 1 or 2 diabetes mellitus and/or hypoglycemia), cardiovascular (including, but not limited to history of myocardial infarction, peripheral arterial disease, stroke), pulmonary (including uncontrolled asthma), hepatic, renal, gastrointestinal, hematologic, immunologic, dermatologic, rheumatic (including gout), and/or biliary, that, in the opinion of the Clinical Investigator (has MD qualifications), could interfere with the interpretation of the study results.
13. Subject has had a loss of 400 mL of blood (e.g., blood/plasma donation) during the prior 30 d of visit 2 (day 0).
14. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
15. Subject has a history of bariatric surgery for weight reducing purposes within the past year.
16. Subject has recently (within 6 months prior to Visit 1; day -7) had a weight loss or gain >4.5 kg.
17. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at Visit 1 (day -7). One re-test will be allowed on a separate day prior to Visit 2 (day 0), for subjects with abnormal blood pressure.
18. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian, ketogenic diet, calorie deprivation), in the opinion of the Clinical Investigator.
19. Subject has used any foods and/or dietary supplements containing medium chain triglycerides (MCT) with 30 d prior to Visit 1 (day -7).
20. Subject has been exposed to any non-registered drug product within 30 d prior to Visit 1 (day -7).
21. Subject has a recent history of (within 12 months of screening; Visit 1; day -7) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
22. Individual has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24
  Area under the curve (AUC) from pre-product consumption (t = -0.25 h) to 24 h (AUC-0.25-24h)
Maximum plasma concentration (Cmax) | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24
Time to Cmax (Tmax) | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24
Elimination rate constant | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24
Half life (t1/2) | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24
Apparent oral clearance (CL/F) | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24

OTHER OUTCOMES:
Adverse Events | Day 2 and Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- BioFortis Innovative Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No